CLINICAL TRIAL: NCT06785038
Title: Encouraging Multiple PrEP Options for Women Engaged in PRimary Care
Acronym: EMPOWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Stacy C Bailey, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STU00220528
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-05

CONDITIONS: PrEP Education
Keywords: PrEP; cisgender women; primary care; electronic health record

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Attention Control (Other)
  Interventions: Behavioral: Attention Control
- EMPOWER Strategy (Experimental)
  Interventions: Behavioral: EMPOWER Strategy

INTERVENTIONS:
Behavioral: EMPOWER Strategy — The EMPOWER Strategy will: 1) identify women in primary care; 2) deliver understandable, actionable, and non-stigmatizing PrEP education, in multiple formats and languages, directly and securely to women via the patient portal; 3) enable women to discreetly self-schedule a visit to discuss PrEP options via the patient portal, with either their own PCP or with a female PCP who has years of experience in PrEP delivery; and 4) support PCP counseling via clinical decision support that provides standardized, patient-centered language to guide PrEP discussions and via 'smart sets' to facilitate PrEP prescribing, when desired and appropriate.
  Other Names: PrEP Education; PrEP Scheduling; PrEP Counseling Support; PrEP Prescribing Support
  Arms: EMPOWER Strategy
Behavioral: Attention Control — Women in this arm will be sent, via the patient portal, a CDC patient education material on benefits of physical activity. The material will be in English or Spanish based on patient's language.
  Arms: Attention Control

SUMMARY:
This study will address the significant yet often overlooked problem of HIV among cisgender women. To do this, researchers will adapt and test a multilingual technology-based strategy supporting informed decision-making for PrEP in primary care. Specifically, researchers will use the electronic health record to securely send women multimedia educational materials in English or Spanish about PrEP, and facilitate electronic scheduling of PrEP visits - if women decide they are interested. Choice is critical.

DETAILED DESCRIPTION:
This study will adapt and pilot test a technology-enabled, primary care-based, health literacy strategy to empower women with increased vulnerability to HIV to make informed decisions about PrEP.

Nearly 20% of new HIV infections in the United States (US) occur among cisgender women, with women of color disproportionately affected. Pre-exposure prophylaxis (PrEP) is a safe, effective, and empowering option for HIV prevention women can initiate and use without partner negotiation. Yet most women are unaware PrEP is an option for them. With primary care representing the frontline of healthcare for most adult women, it is an ideal setting to promote PrEP awareness and informed decision-making. Importantly, women themselves have asked for PrEP discussions to be normalized in primary care and multiple studies have shown that women value talking with clinicians about PrEP. Unfortunately, many primary care providers (PCPs) lack the time, resources, and experience needed to counsel women on PrEP during busy, routine visits. Our proposed R34 Encouraging Multiple PrEP Options for Women Engaged in PRimary Care (EMPOWER) therefore offers a pragmatic and innovative approach to the delivery of PrEP information to women in primary care. The EMPOWER strategy addresses well-documented barriers and 'missed opportunities' for HIV prevention among cisgender women and supports informed PrEP decision-making by: 1) identifying women in primary care; 2) delivering understandable, actionable, and non-stigmatizing PrEP education, in multiple formats and languages, directly and securely to women via the patient portal; 3) enabling women to discreetly self-schedule a visit to discuss PrEP options with either their own PCP or with a female PCP who has years of experience in PrEP delivery; and 4) supporting PCP counseling via clinical decision support that provides standardized, patient-centered language to guide PrEP discussions and 'smart sets' to facilitate PrEP prescribing, when desired. Our specific aims are to: 1) Adapt and coordinate the EMPOWER strategy to support informed decision-making among diverse cisgender women with increased vulnerability to HIV seen in primary care; 2) Pilot test the efficacy of the EMPOWER strategy, compared to an attention control, on PrEP knowledge, stigma, and future intention to use PrEP; and 3) Assess the reach, adoption, implementation, and maintenance of EMPOWER components. EMPOWER will be evaluated in Cook County, an 'Ending the HIV Epidemic' priority area. The study will be meaningfully informed by a community advisory board of diverse women, a scientific advisory board of clinicians and experts, and a community collaboration board of local organization leaders in the field of HIV.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

* identify as a cisgender woman
* be aged 18 years or older
* speak English or Spanish
* be a primary care patient at the participating health center
* have an active patient portal account
* be HIV negative
* have never been prescribed PrEP

Exclusion Criteria:

Individuals will be excluded if they have any:

- severe, uncorrectable vision, hearing, or cognitive impairments that would preclude study consent or participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender women
Enrollment: 120 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
PrEP Knowledge | Two to 4 weeks after women are sent materials (attention control or EMPOWER Strategy) in their patient portal accounts
  PrEP knowledge is our primary outcome. We will use an adapted version of an existing PrEP knowledge scale by Walsh (2019). Participants will be asked 13 questions, each with true, false or don't know response options. The number of correct answers will be summed and expressed as percentage correct. Higher scores will represent greater PrEP knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy C Bailey, PhD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
All IDP collected throughout the trial will be included.
Supporting Information: SAP
Time Frame: April 2026 for at least 3 years
Access Criteria: We will submit de-identified data to the NIMH Data Archive.
URL: https://nda.nih.gov/